CLINICAL TRIAL: NCT06504394
Title: A Phase 2 Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Subcutaneous Pembrolizumab Coformulated With Hyaluronidase (MK-3475A) in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma (rrcHL) or Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
Brief Title: A Study to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) Coformulated With Berahyaluronidase Alfa (MK-3475A) in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma (rrcHL) or Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)(MK-3475A-F65)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-F65; MK-3475A-065 (Other: MSD); 2024-510969-42-00 (Registry Identifier: EU CT); U1111-1302-8349 (Registry Identifier: UTN)
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Classical Hodgkin Lymphoma Recurrent; Classical Hodgkin Lymphoma Refractory; Primary Mediastinal Large B-cell Lymphoma Recurrent; Primary Mediastinal Large B-cell Lymphoma Refractory
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death-2 (PD2, PD-2); Programmed Death-Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Coformulated With Hyaluronidase (Experimental): Participants with rrCHL and rrPMBCL receive pembrolizumab coformulated with hyaluronidase subcutaneous (SC) injection on Day 1 of each 6-week cycle (Q6W) for up to 18 cycles (approximately 2 years) until documented disease progression per investigator assessment.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — SC injection
  Other Names: MK-3475A

SUMMARY:
The primary purpose of the study is to assess the pharmacokinetics (PK) profile of pembrolizumab following subcutaneous (SC) injection of pembrolizumab coformulated with hyaluronidase, and to evaluate the objective response rate (ORR) of pembrolizumab (+) berahyaluronidase alfa SC in adult participants with Relapsed or Refractory Classical Hodgkin Lymphoma (rrcHL) or Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL). There is no formal hypothesis to be tested for this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically confirmed diagnosis of classical Hodgkin lymphoma (cHL) or primary mediastinal B-cell lymphoma (PMBCL)
* Radiographically measurable cHL or PMBCL disease assessed by investigator as per Lugano classification
* Have a life expectancy of >3 months
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load before enrollment
* Participants with history of hepatitis C virus (HCV) infection are eligible if they have completed curative antiviral therapy at least 4 weeks before enrollment and HCV viral load is undetectable at screening
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before or on the day of the first dose of study intervention

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has clinically significant (i.e., active) cardiovascular disease
* Has pericardial effusion or clinically significant pleural effusion
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Received prior monoclonal antibody within 4 weeks prior to first dose of study intervention or has not recovered (i.e., ≤Grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti-PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before first dose of study intervention
* Is receiving systemic antineoplastic chemotherapy, immunotherapy, or biological therapy not specified in this protocol
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy except certain protocol-specified therapies
* Concurrent active hepatitis B and hepatitis C virus infection
* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic stem cell transplant (SCT) within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2028-11-08 (Estimated); Study Completion 2028-11-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Lugano Classification Criteria as Assessed by Investigator | Up to approximately 48 months
  ORR is defined as the percentage of the participants who had complete response (CR) or partial response (PR) and will be evaluated using computed tomography (CT) and positron emission tomography (PET)-CT. Response was assessed based on the International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants who experience CR or PR as assessed by investigator will be presented.
Maximum Concentration (Cmax) of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of Cmax. Cmax is defined as the peak concentration of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase.
Lowest Plasma Concentration (Ctrough) of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of Ctrough. Ctrough is defined as the lowest concentration of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase.
Area Under the Concentration-Time Curve of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase from Week 0-Week 6 (AUC0-6weeks) | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of AUC0-6weeks. AUC0-6 weeks is defined as area under concentration time curve over a 6-week dosing interval of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase.

SECONDARY OUTCOMES:
Duration of Response (DOR) per Lugano Classification Criteria as Assessed by Investigator | Up to approximately 48 months
  For participants who demonstrate a confirmed complete response (CR) or partial response (PR), DOR is defined as the time from CR or PR to documented disease progression or death. Participants are assessed using computed tomography (CT) and positron emission tomography (PET)-CT and response was evaluated based on the Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). CR is complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters (SPD) for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR as assessed by the investigator will be presented.
Number of Participants with Antidrug Antibodies (ADA) Level of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase | At designated timepoints (Up to approximately 27 months)
  Blood samples will be collected at designated time points for the determination of the presence or absence of ADA of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase. The number of participants who develop ADA will be reported.
Maximum Concentration (Cmax) of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase at Steady-State | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of Cmax. Cmax is defined as the peak concentration of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase at steady-state.
Lowest Plasma Concentration (Ctrough) of Pembrolizumab After Administration of SC Pembrolizumab Coformulated with Hyaluronidase at Steady-State | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of Ctrough. Ctrough is defined as the lowest concentration of pembrolizumab after administration of SC pembrolizumab coformulated with hyaluronidase at steady-state.
Area Under the Concentration-Time Curve of Pembrolizumab After Administration of SC Pembrolizumab coformulated with Hyaluronidase from Week 0-Week 6 (AUC0-6weeks) at Steady-State | At designated time points (up to ~6 weeks)
  Blood samples will be collected at designated timepoints for the determination of AUC0-6weeks. AUC0-6 weeks is defined as area under concentration time curve over a 6-week dosing interval of pembrolizumab coformulated with hyaluronidase at steady-state.
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 30 months
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of participants who experience an AE will be reported.
Number of Participants Discontinuing Study Treatment due to an Adverse Event (AE) | Up to approximately 2 years
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- United States (4):
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 0115), Iowa City, Iowa
  - University of Iowa - Waukee ( Site 0111), Waukee, Iowa
  - Comprehensive Cancer Centers of Nevada ( Site 0114), Las Vegas, Nevada
  - Clinical Research Alliance ( Site 0101), Westbury, New York
- Westmead Hospital ( Site 0901), Westmead, New South Wales, Australia
- Chile (5):
  - IC La Serena Research ( Site 0204), La Serena, Coquimbo Region
  - FALP ( Site 0207), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 0201), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0202), Santiago, Region M. de Santiago
  - Biocenter ( Site 0203), Concepción, Región del Biobío
- Universitaetsklinikum Essen ( Site 1302), Essen, North Rhine-Westphalia, Germany
- Mexico (2):
  - Health Pharma Professional Research S.A. de C.V: ( Site 0403), Mexico City, Mexico City
  - Centro de Investigacion Clinica de Oaxaca ( Site 0405), Oaxaca City
- Auckland City Hospital ( Site 1001), Auckland, New Zealand
- Poland (4):
  - Pratia MCM Krakow ( Site 0503), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Kilinka Onkologii I Hematologii ( Site 0501), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 0502), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0504), Gliwice, Silesian Voivodeship
- Seoul National University Hospital-Oncology ( Site 1101), Seoul, South Korea
- Spain (3):
  - Institut Català d'Oncologia - L'Hospitalet-Haematology Department ( Site 0703), L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario de Salamanca ( Site 0702), Salamanca, Castille and León
  - Hospital Universitario 12 de Octubre-Hemathology and hemotherapy ( Site 0701), Madrid
- Turkey (Türkiye) (3):
  - Ankara Universitesi Tıp Fakultesi Hastanesi ( Site 0801), Ankara
  - Hacettepe Universite Hastaneleri ( Site 0802), Ankara
  - Ondokuz Mayıs Universitesi ( Site 0803), Samsun
- United Kingdom (4):
  - Glan Clwyd Hospital ( Site 0602), Bodelwyddan, Denbighshire
  - University College London Hospital ( Site 0605), London, London, City of
  - Churchill Hospital ( Site 0604), Oxford, Oxfordshire
  - The Christie NHS Foundation Trust ( Site 0603), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26323&tenant=MT_MSD_9011